CLINICAL TRIAL: NCT03635229
Title: Risk Factor of Postoperative Delirium and Postoperative Cognitive Decline After Cardiac Surgery
Brief Title: Risk Factor of POD and POCD After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 705/2560(EC1)
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction
Keywords: cardiac surgery; perioperative care; postoperative delirium; postoperative cognitive dysfunction
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative delirium (POD) and postoperative cognitive decline (POCD) are common after surgeries in the elderly, especially after cardiothoracic surgery. These conditions are associated with adverse short- and long-term outcomes.

Multiple conditions in the perioperative period have been proposed as risk factors of POD and POCD.

Incidences vary across institutions due to differences in screening and diagnostic tools.

DETAILED DESCRIPTION:
This is a prospective observational study to identify the incidences and risk factors of postoperative delirium and postoperative cognitive decline after elderly patients undergoing cardiac surgical procedures which require cardiopulmonary bypass and postoperative intensive care unit (ICU) admission.

Patients will be screen for POD and POCD with various psychological tests in the postoperative period and after hospital discharge.

Perioperative data and outcomes will be used to identify risk factors of both conditions.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years old or older
* undergoing open heart surgery (cardiopulmonary bypass assisted cardiothoracic surgery

Exclusion Criteria:

* unable to communicate
* severe visual or hearing impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients (age 65 and older) undergoing cardiopulmonary bypass- assisted surgery with anticipated postoperative intensive care unit admission
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2018-08-21 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | Postoperative day 1-5 (5 consecutive days)
  A result consistent with postoperative delirium by using Confusion Assessment Method-ICU (CAM-ICU) in the postoperative period

SECONDARY OUTCOMES:
Postoperative cognitive dysfunction - postoperative | Postoperative day 5-9 (5 consecutive days)
  A result consistent with postoperative cognitive dysfunction by using Montreal Cognitive Assessment (MOCA)
Postoperative cognitive dysfunction - 3 month | At 3rd month after hospital discharge
  A result consistent with postoperative cognitive dysfunction by using Montreal Cognitive Assessment (MOCA)
Postoperative cognitive dysfunction - 1 year | At 12th month after hospital discharge
  A result consistent with postoperative cognitive dysfunction by using Montreal Cognitive Assessment (MOCA)

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No